CLINICAL TRIAL: NCT04810091
Title: TELEHEART: Telotristat Ethyl in a Heart Biomarker Study
Brief Title: Telotristat Ethyl for the Treatment of Carcinoid Heart Disease in Patients With Metastatic Neuroendocrine Tumor
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1205; NCI-2021-00852 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1205 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-03-04; First posted 2021-03-22 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Neuroendocrine Neoplasm; Metastatic Neuroendocrine Neoplasm
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — telotristat ethyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (telotristat ethyl, SSA) (Experimental): Patients receive telotristat ethyl PO TID and SSA for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Questionnaire Administration; Drug: Telotristat Ethyl
- Arm B (placebo, SSA) (Active Comparator): Patients receive placebo PO TID and SSA for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Placebo Administration — Given PO
  Arms: Arm B (placebo, SSA)
Other: Questionnaire Administration — Ancillary studies
Drug: Telotristat Ethyl — Given PO
  Arms: Arm A (telotristat ethyl, SSA)

SUMMARY:
This phase III trial compares the effect of telotristat ethyl and the current standard of care somatostatin analog therapy or somatostatin analog therapy alone in treating patients with neuroendocrine tumor that has spread to other places in the body (metastatic). Telotristat ethyl and somatostatin analog therapy may help to control carcinoid syndrome and carcinoid heart disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the percent change in N-terminal pro B-type natriuretic peptide (NT-proBNP) at 6 month visit from baseline after initiation of study drug in each arm and to compare the percent change between the two study arms.

SECONDARY OBJECTIVES:

I. To evaluate the change in functional capacity from baseline at 3 and 6 month visits as assessed by a 6 minute walk test (6MWT) in each arm.

II. To evaluate changes in echocardiographic parameters (Carcinoid Valvular Heart Disease [CVHD] score, global longitudinal myocardial strain assessment of the left and right ventricle/tricuspid annular plane systolic excursion [TAPSE]) from baseline to 3 and 6 month visits in each arm.

III. To evaluate the change from baseline to 3 and 6 month visits in plasma 5-hydroxyindoleacetic acid (5-HIAA) levels in each arm.

IV. To evaluate the change from baseline to 3 and 6 month visits in high sensitivity troponin T in each arm.

V. To evaluate the change from baseline to 3 and 6 month visits in health related quality of life with using the MD Anderson Symptom Inventory (MDASI) in each arm.

VI. To evaluate compliance of medications.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive telotristat ethyl orally (PO) three times daily (TID) and somatostatin analog therapy (SSA) for 6 months in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive placebo PO TID and SSA for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are >= 18 years old will be eligible for the study
* Histopathologically-confirmed,metastatic neuroendocrine tumor and/or locally/regionally advanced neuroendocrine tumor
* Documented history of carcinoid syndrome based on clinical parameters
* Currently receiving stable-dose somatostatin analog (SSA) therapy defined as >= 2 months

  * Dose of long-acting release (LAR) or depot SSA therapy and on at least:

    * Octreotide LAR at 30 mg every 4 weeks
    * Lanreotide depot at 120 mg every 4 weeks
    * Patients who cannot tolerate SSA therapy at a level indicated above will be allowed to enter at their highest tolerated dose
* Ability and willingness to provide written informed consent
* Patients of childbearing potential must agree to use an adequate method of contraception during the study and for 30 days after the last dose of telotristat ethyl

  * Childbearing potential is defined as those who have not undergone surgical sterilization (eg. documented hysterectomy, tubal ligation, or bilateral salpingo-oophorectomy) or those who are not considered postmenopausal (defined as 12 months of spontaneous amenorrhea).
  * Adequate methods of contraception, defined as having a failure rate of < 1% per year, for patients or their partner include the following: condom with spermicidal gel, diaphragm with spermicidal gel, intrauterine device, surgical sterilization, vasectomy, oral contraceptive pill, depo-progesterone injections, progesterone implant (ie, Implanon), patch (Ortho Evra), NuvaRing, and abstinence. If a patient is not sexually active but becomes active, he or his partner should use medically accepted forms of contraception
* Eastern Cooperative Oncology Group (ECOG) 0-2

Exclusion Criteria:

* Previous exposure to telotristat ethyl (XERMELO) in the last 3 months
* History of active treatment for malignancy, other than neuroendocrine tumor (malignancies that in the opinion of the Investigator are considered cured, may participate)
* Treatment with any tumor directed therapy, including interferon, chemotherapy, mechanistic target of rapamycin (mTOR) inhibitors < 4 weeks prior to screening, or hepatic embolization, radiotherapy, peptide receptor radionuclide therapy, and/or tumor debulking < 12 weeks prior to screening
* History of short bowel syndrome or other known causes of diarrhea unrelated to carcinoid syndrome
* Clinically significant (as per primary investigators judgement) cardiac arrhythmia, bradycardia, tachycardia that would compromise patient safety or the outcome of the study
* Estimated glomerular filtration rate estimated glomerular filtration rate (eGFR) < 30 ml/min
* Hepatic laboratory values of aspartate transaminase (AST) or alanine aminotransferase (ALT):

  * > 5 x upper limit of normal (ULN) if patient has documented history of hepatic metastases; or
  * > 2.5 x ULN if no liver metastases are present
* Pregnant or lactating patients
* Patients receiving everolimus due to poor response to SSA
* Life expectancy < 6 months
* Any other clinically significant laboratory abnormality that would compromise patient safety or the outcome of the study as per primary investigators judgement
* Any clinically significant and/or uncontrolled cardiac-related abnormality that would compromise patient safety or the outcome of the study including as per primary investigators judgement, but not limited to:

  * Arrhythmia causing hemodynamic compromise
  * Symptomatic severe valvular disease
  * Symptomatic congestive heart failure classified by New York Heart Association (NYHA) class IV
  * Evidence of ischemia on electrocardiography (ECG) with chest pain
  * Unstable angina pectoris
* Current complaints of persistent constipation or history of chronic constipation, bowel obstruction or fecaloma within the past 6 months
* Investigator assessment of known history and/or uncontrolled hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus (HIV)-1 or HIV-2
* History of substance or alcohol abuse (Diagnostic and Statistical Manual of Mental Disorders 5th edition [DSM-V] Criteria for Substance-Related Disorders) within the past 2 years
* History of galactose intolerance, deficiency of Lapp lactase, or glucose-galactose malabsorption
* Receipt of any investigational agent or study treatment (other treatment nor approved by Food and Drug Administration [FDA] for carcinoid syndrome or carcinoid heart disease) within the past 30 days
* Existence of any surgical or medical condition that, in the judgment of the Investigator, might compromise patient safety or the outcome of the study
* Presence of any clinically significant findings (relative to the patient population) during review of medical history or upon PE that, in the investigator's opinion, would compromise patient safety or the outcome of the study (e.g., psychiatric illness/social situations that would limit compliance with study requirements)
* Unable or unwilling to communicate or cooperate with the Investigator for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-08-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cezar A Iliescu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 79 participants who consented and enrolled in the study, 6 withdrew before arm assignment. These 6 participants were not randomized and were excluded from the study. The remaining 73 participants were randomized to one of two arms.
Groups:
- Placebo + SSA: Placebo-matching telotristat ethyl tablet TID + stable-dose somatostatin analog (SSA) therapy
- Xermelo + SSA: Telotristat ethyl 500 mg po TID + stable-dose somatostatin analog (SSA)
Period: Overall Study
Arm/Group | Placebo + SSA | Xermelo + SSA
Started | 37 | 36
Randomized | 37 | 36
Treated | 35 | 32
3 Month Follow-up | 29 | 29
Completed | 27 | 26
Not Completed | 10 | 10
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Ineligible | 0 | 1
Not completed — Non-compliance | 0 | 1
Not completed — Prescribed Xermelo by local oncologist | 1 | 0
Not completed — Progressive disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + SSA | Xermelo + SSA | Total
Number analyzed (Participants) | 37 | 36 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 42
  >=65 years | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (11.6) | 59.2 (14.4) | 61.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 23 | 20 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 32 | 29 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 37 | 36 | 73

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in NTproBNP at 6 Months Visit From Baseline
Description: Percent change in N-terminal pro B-type natriuretic peptide (NT-proBNP) from baseline to 6 months defined as (NTproBNP at 6 month - NTproBNP at baseline)/(NTproBNP at baseline)*100
Time Frame: Baseline and at 6 months
Population: Patients who had NTproBNP at both baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 27 | 26
Percent change from baseline | -9.1 [-32.4 to 14.3] | 1.4 [-32.4 to 53.8]

2. Secondary Outcome: Change in 6MWT at 3 Month Visit
Description: Change in functional capacity from baseline to 3-month visit, assessed by a 6-minute walk test (6MWT), where 6MWT is defined as the distance walked in 6 minutes, and the change is calculated as: 6MWT at 3 months minus 6MWT at baseline
Time Frame: Baseline and 3 month follow-up
Population: Of the 29 participants who completed 3-month follow-up in the Placebo + SSA arm, 25 completed the 6MWT at both baseline and 3 months. In the Xermelo + SSA arm, all 29 participants who completed 3-month follow-up also completed the 6MWT at both baseline and at 3 months.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 25 | 29
meters | 0 [-35 to 45] | 8 [-25 to 64]

3. Secondary Outcome: Change in 6MWT at 6 Month Visit
Description: Change in functional capacity from baseline to 6-month visit, assessed by a 6-minute walk test (6MWT), where 6MWT is defined as the distance walked in 6 minutes, and the change is calculated as: 6MWT at 6 months minus 6MWT at baseline
Time Frame: Baseline and 6 month follow-up
Population: Of the 27 participants who completed 6-month follow-up in the Placebo + SSA arm, 26 participants completed 6MWT at both baseline and at 6 months. All 26 participants who completed 6-month follow-up in the Xermelo + SSA arm completed the 6MWT at both baseline and 6 months.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 26 | 26
meters | -14 [-63 to 39] | 25.5 [-27 to 67]

4. Secondary Outcome: Change in CVHD % Score From Baseline to 3 Month Visit
Description: The Carcinoid Valvular Heart disease (CVHD) % score at 3 months minus CVHD % score at baseline. CVHD score was determined by 1) tricuspid valve appearance, 2) tricuspid regurgitation severity by either spectral pulsed wave or color dopplet flow mapping, 3) pulmonary stenosis severity by spectral pulsed or continuous wave Doppler, and 4) pulmonary insufficiency severity by color Doppler. CVHD % score was calculated as total points assigned across four echo parameters (specified above 1-4)) divided by the maximum possible points (14) and multiplied by 100. The CVHD % score ranges from 0% to 100%, with higher values indicating more severe disease. The change in CVHD % score from baseline to 3 months reflects disease progression or improvement: a positive change indicates worsening valvular involvement, a negative change indicates improvement, and zero indicates stability.
Time Frame: Baseline and 3 month follow-up
Population: Of the 29 participants who completed 3-month follow-up in the Placebo + SSA arm, 7 completed CVHD evaluations at both baseline and 3 months. In the Xermelo + SSA arm, 5 of the 29 participants who completed 3-month follow-up completed CVHD evaluations at both baseline and 3 months.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 7 | 5
Scores on a scale | 0 [-7 to 0] | 0 [0 to 0]

5. Secondary Outcome: Change in CVHD Score From Baseline to 6 Month Visit
Description: The Carcinoid Valvular Heart disease (CVHD) % score at 6 months minus CVHD % score at baseline. CVHD score was determined by 1) tricuspid valve appearance, 2) tricuspid regurgitation severity by either spectral pulsed wave or color dopplet flow mapping, 3) pulmonary stenosis severity by spectral pulsed or continuous wave Doppler, and 4) pulmonary insufficiency severity by color Doppler. CVHD % score was calculated as total points assigned across four echo parameters divided by the maximum possible points (14) and multiplied by 100. The CVHD % score ranges from 0% to 100%, with higher values indicating more severe disease. The change in CVHD % score from baseline to 6 months reflects disease progression or improvement: a positive change indicates worsening valvular involvement, a negative change indicates improvement, and zero indicates stability.
Time Frame: Baseline and 6 month follow-up
Population: Of the 27 participants who completed 6-month follow-up in the Placebo + SSA arm, 24 participants completed CVHD evaluations at both baseline and 6 months. In the Xermelo + SSA arm, 23 of the 26 participants who completed 6-month follow-up completed CVHD evaluation at both baseline and at 6 months. The values reported represent the median values for change in CVHD score for each Arm, and do not represent non-meaningful placeholders.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 24 | 23
Scores on a scale | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Percentage of Participants With Significant Change in Strain-RV From Baseline at 3 Months
Description: Percentage of participants with a significant change in right ventricular global longitudinal strain (strain-RV) from baseline to 3 months. A significant change is defined as an 15% or more change (increase or decrease) from baseline to 3 months. The Exact 2-sided 95% CI is based on the observed proportion of participants.
Time Frame: Baseline and 3 month follow-up
Population: Of the 29 participants who completed 3 months follow-up in the Placebo + SSA arm, 3 completed strain RV evaluations at both baseline and 3 months. In the Xermelo + SSA arm, 7 of the 29 participants who completed 3-month follow-up completed strain RV evaluations at both baseline and at 3 months.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 3 | 7
Percentage of Participants | 33.3 [0.8 to 90.6] | 42.9 [9.9 to 81.6]

7. Secondary Outcome: Percentage of Participants With Significant Change in Strain-RV From Baseline at 6 Months
Description: Percentage of participants with a significant change in right ventricular global longitudinal strain (strain-RV) from baseline to 6 months. A significant change is defined as an 15% or more change (increase or decrease) from baseline to 6 months. The Exact 2-sided 95% CI is based on the observed proportion of participants.
Time Frame: Baseline and 6 month follow-up
Population: Of the 27 participants who completed 6-month follow-up in the Placebo + SSA arm, 7 completed strain RV evaluations at both baseline and 6 months. In the Xermelo + SSA arm, 5 of the 26 participants who completed 6-month follow-up completed strain RV evaluations at both baseline and 6 months.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 7 | 5
Percentage of Participants | 42.9 [9.9 to 81.6] | 40 [5.3 to 85.3]

8. Secondary Outcome: Percentage of Participants With Significant Change in Strain-LV From Baseline at 3 Months
Description: Percentage of participants with a significant change in left ventricular global longitudinal strain (strain-LV) from baseline to 3 months. A significant change is defined as an 15% or more change (increase or decrease) from baseline to 3 months. The Exact 2-sided 95% CI is based on the observed proportion of participants.
Time Frame: Baseline and 3 month follow-up
Population: Of the 29 participants who completed 3-month follow-up in the Placebo + SSA arm, 7 participants completed strain LV evaluations at both baseline and 3 months. In the Xermelo + SSA arm, 7 of the 29 participants who completed 3-month follow-up completed strain LV evaluations at both baseline and 3 months.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 7 | 7
Percentage of Participants | 14.3 [0.4 to 57.9] | 28.6 [3.7 to 71.0]

9. Secondary Outcome: Percentage of Participants With Significant Change in Strain-LV From Baseline at 6 Months
Description: Percentage of participants with a significant change in left ventricular global longitudinal strain (strain-LV) from baseline to 6 months. A significant change is defined as an 15% or more change (increase or decrease) from baseline to 6 months. The Exact 2-sided 95% CI is based on the observed proportion of participants.
Time Frame: Baseline and 6 month follow-up
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 15 | 16
Percentage of Participants | 13.3 [1.7 to 40.5] | 12.5 [1.6 to 38.4]

10. Secondary Outcome: Percentage of Participants With Normal TAPSE at 3 Months
Description: Percentage of participants with a normal Tricuspid Annular Plane Systolic Excursion (TAPSE) at 3 months, where TAPSE ≥1.6cm is defined as normal. The Exact 2-sided 95% CI is based on the observed proportion of participants.
Time Frame: 3 month follow-up
Population: Among 29 who completed 3 months follow-up in the Placebo + SSA arm, 5 participants completed TAPSE evaluations at both baseline and at 3 months. In the Xermelo + SSA arm, 7 of the 29 participants who completed TAPSE evaluations at both baseline and at 3 months.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 5 | 7
Percentage of Participants | 100 [47.8 to 100] | 86 [42.1 to 99.6]

11. Secondary Outcome: Percentage of Participants With Normal TAPSE at 6 Months
Description: Percentage of participants with a normal Tricuspid Annular Plane Systolic Excursion (TAPSE) at 6 months, where TAPSE ≥1.6cm is defined as normal. The Exact 2-sided 95% CI is based on the observed proportion of participants.
Time Frame: 6 month follow-up
Population: Of the 27 participants who completed 6-month follow-up in the Placebo + SSA arm, 21 completed TAPSE evaluations at both baseline and 6 months. In Xermelo + SSA arm, 20 of the 26 who completed 6-month follow-up ccompleted TAPSE evaluation at both baseline and 6 months.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 21 | 20
Percentage of Participants | 100 [83.9 to 100] | 95 [75.1 to 99.9]

12. Secondary Outcome: Change in 5HIAA From Baseline to 3 Months
Description: Change in plasma 5HIAA (5-Hydroxyindoleacetic acid) level from baseline to 3 months. The change is calculated as: 5HIAA at 3 months minus 5HIAA at baseline
Time Frame: Baseline and 3 month follow-up
Population: Of the 29 participants who completed 3-month follow-up in the Placebo + SSA arm, 26 completed 5HIAA evaluations at both baseline and 3 months. In Xermelo + SSA arm, all 29 who completed 3-month follow-up completed 5HIAA evaluations at both baseline and 3 months.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 26 | 29
ng/mL | -0.9 [-4.2 to 6.6] | -55.3 [-118.2 to -28.6]

13. Secondary Outcome: Change in 5HIAA From Baseline to 6 Months
Description: Change in 5HIAA measurement from baseline to 6 months
Time Frame: Baseline and 6 month follow-up
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 26 | 26
ng/mL | 0.1 [-1.9 to 7.3] | -56.4 [-104.4 to -18.6]

14. Secondary Outcome: Change in Troponin From Baseline to 3 Months
Description: Change in troponin level from baseline to 3 months, calculated as: troponine at 3 months minus troponin at baseline
Time Frame: Baseline and 3 months follow-up
Population: Of the 29 participants who completed 3-month follow-up in the Placebo + SSA arm, 25 completed troponin evaluation at both baseline and 3 months. In the Xermelo + SSA arm, 25 of the 29 who completed 3-month completed troponin evaluation at both baseline and 3 months.
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 25 | 25
ng/L | 0 [-1 to 2] | 0 [-2 to 1]

15. Secondary Outcome: Change in Troponin From Baseline to 6 Months
Description: Change in troponin level from baseline to 6 months, calculated as: troponine at 6 months minus troponin at baseline
Time Frame: Baseline and 6 months follow-up
Population: Of the 27 participants who completed 6-month follow-up in the Placebo + SSA arm, 26 completed troponin evaluation at both baseline and 6 months. In the Xermelo + SSA arm, 25 of the 26 who completed 6-month follow-up completed troponin evaluation at both baseline and at 6 months.
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 26 | 25
ng/L | 0 [-1 to 1] | 0 [-2 to 1]

16. Secondary Outcome: Change in MDASI Mean Core Symptom Score From Baseline to 3 Months
Description: Change in MD Anderson Symptom Inventory (MDASI) mean core symptom score from baseline to 3 months. The MDASI mean core symptom score is calculated as the mean of 13 core symptom items, each ranged from 0 ( "not present") to 10 being ("as bad as you can imagine"), with the higher scores indicating worse symptoms. The change is computed as: score at 3 months minus score at baseline
Time Frame: Baseline and 3 months follow-up
Population: Of the 29 participants who completed 3-month follow-up in the Placebo + SSA arm, 27 completed MDASI core symptom evaluation at both baseline and 3 months. In the Xermelo + SSA arm, 28 of the 29 participants who completed 3-month follow-up completed MDASI core symptom evaluation at both baseline and 3 months.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 27 | 28
Scores on a scale | -0.2 [-0.4 to 0.4] | 0.1 [-0.2 to 0.3]

17. Secondary Outcome: Change in Core Symptom Score From Baseline to 6 Months
Description: Change in MD Anderson Symptom Inventory (MDASI) mean core symptom score from baseline to 6 months. The MDASI mean core symptom score is calculated as the mean of 13 core symptom items, each ranged from 0 ( "not present") to 10 being ("as bad as you can imagine"), with the higher scores indicating worse symptoms. The change is computed as: score at 6 months minus score at baseline
Time Frame: Baseline and 6 months follow-up
Population: All 27 participants who completed 6-month follow-up in the Placebo + SSA arm completed MDASI core symptom evaluation at both baseline and 6 months. In the Xermelo + SSA arm, 25 of the 26 participants who completed 6-month follow-up completed MDASI core symptom evaluation at both baseline and 6 months.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 27 | 25
Scores on a scale | 0 [-0.3 to 0.4] | 0 [-0.3 to 0.2]

18. Secondary Outcome: Change in MDASI Mean Total Symptom Score From Baseline to 3 Months
Description: Change in MD Anderson Symptom Inventory (MDASI) mean total symptom score from baseline to 3 months. The MDASI mean total symptom score is calculated as the mean symptom severity of 21 symptom items (13 core symptom items and 8 additional symptom items), each ranged from 0 ( "not present") to 10 being ("as bad as you can imagine), with the higher scores indicating worse symptoms. The change is computed as: score at 3 months minus score at baseline
Time Frame: Baseline and 3 months follow-up
Population: Of the 29 participants who completed 3-month follow-up in the Placebo + SSA arm, 27 completed MDASI total symptom evaluation at both baseline and 3 months. In the Xermelo + SSA arm, all 28 participants who completed 3-month follow-up completed MDASI total symptom evaluation at both baseline and 3 months.
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 27 | 28
points | 0 [-0.3 to 0.5] | 0 [-0.2 to 0.2]

19. Secondary Outcome: Change in MDASI Mean Total Symptom Score From Baseline to 6 Months
Description: Change in MD Anderson Symptom Inventory (MDASI) mean total symptom score from baseline to 6 months. The MDASI mean total symptom score is calculated as the mean symptom severity of 21 symptom items (13 core symptom items and 8 additional symptom items), each ranged from 0 ( "not present") to 10 being ("as bad as you can imagine), with the higher scores indicating worse symptoms. The change is computed as: score at 6 months minus score at baseline
Time Frame: Baseline and 6 months follow-up
Population: All 27 participants who completed 6-month follow-up in the Placebo + SSA arm completed MDASI total symptom evaluation at both baseline and 6 months. In the Xermelo + SSA arm, 25 of the 26 participants who completed 6-month follow-up completed MDASI total symptom evaluation at both baseline and 6 months.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 27 | 25
Scores on a scale | -0.1 [-0.2 to 0.2] | 0 [-0.4 to 0.3]

20. Secondary Outcome: Change in MDASI Mean Interference Score From Baseline to 3 Months
Description: Change in MD Anderson Symptom Inventory (MDASI) mean interference score from baseline to 3 months. The MDASI mean interference score is calculated as the mean of 6 interference items, each ranged from 0 ( "not present") to 10 being ("as bad as you can imagine"), with the higher scores indicating worse interference. The change is computed as: score at 3 months minus score at baseline
Time Frame: Baseline and 3 months follow-up
Population: Of the 29 participants who completed 3-month follow-up in the Placebo + SSA arm, 26 completed MDASI interference evaluation at both baseline and 3 months. In the Xermelo + SSA arm, 28 of the 29 participants who completed 3-month follow-up completed MDASI interference evaluation at both baseline and 3 months.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 26 | 28
Scores on a scale | 0 [-0.3 to 0.8] | 0 [-0.4 to 0.1]

21. Secondary Outcome: Change in Interference Score From Baseline to 6 Months
Description: Change in MD Anderson Symptom Inventory (MDASI) mean interference score from baseline to 6 months. The MDASI mean interference score is calculated as the mean of 6 interference items, each ranged from 0 ( "not present") to 10 being ("as bad as you can imagine"), with the higher scores indicating worse interference. The change is computed as: score at 6 months minus score at baseline
Time Frame: Baseline and 6 months follow-up
Population: Of the 27 participants who completed 6-month follow-up in the Placebo + SSA arm, 26 completed MDASI interferemce evaluation at both baseline and 6 months. In the Xermelo + SSA arm, 24 of the 26 who completed 6-month follow-up completed MDASI interference evaluation at both baseline and 6 months.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 26 | 24
Scores on a scale | 0 [-0.3 to 0.5] | 0 [-0.5 to 0]

22. Secondary Outcome: Compliance>=70% While the Patients Were in the Study
Description: Percentage of participants classified as compliant (compliance≥70%) during the study. Compliance is calculated as the total number of pills taken divided by the toal number of pills dispensed while the patient was on the study. Participants with compliance≥70% are considered compliant; otherwise, not compliant.
Time Frame: Baseline, 3 months follow-up, 6 months follow-up
Population: Those who were treated: 35 in placebo + SSA and 32 in Xermelo + SSA
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo + SSA | Xermelo + SSA
Number analyzed (Participants) | 35 | 32
Percentage of Participants | 74.3 [56.7 to 87.5] | 87.5 [71.0 to 96.5]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline throughout the follow-up period (3-month and 6-month follow-up visits) and for up to 30 days after the last dose of the study drug, with the treatment period planned for 6-months
Arm/Group | Placebo + SSA | Xermelo + SSA
All-Cause Mortality (participants affected / at risk) | 1/35 | 0/32
Serious Adverse Events (participants affected / at risk) | 3/35 | 4/32
Other Adverse Events (participants affected / at risk) | 26/35 | 27/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + SSA (N=35) | Xermelo + SSA (N=32)
Ascites (death) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cataract (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ejection fraction decreased (Cardiac disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + SSA (N=35) | Xermelo + SSA (N=32)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (13) | 20 (21)
Nausea (Gastrointestinal disorders) | 6 (11) | 7 (8)
Constipation (Gastrointestinal disorders) | 5 (6) | 8 (8)
Alkaline phosphtase increased (Investigations) | 3 (4) | 8 (8)
Fatigue (General disorders) | 4 (6) | 5 (5)
Headache (Nervous system disorders) | 4 (5) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
Creatinine increased (Renal and urinary disorders) | 8 (8) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Heart failure (Cardiac disorders) | 1 (1) | 7 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 4 (5)
Cardiac troponin T increased (Investigations) | 1 (1) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1)
Bloating (Gastrointestinal disorders) | 4 (5) | 1 (1)
Edema limbs (General disorders) | 6 (6) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Chest pain - cardiac (Cardiac disorders) | 3 (4) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Flushing (Vascular disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT04810091/Prot_SAP_001.pdf